CLINICAL TRIAL: NCT00595946
Title: A Multi-center, Randomized, Double-Blinded Study of the Efficacy and Safety of Lubiprostone in Patients With Opioid-induced Bowel Dysfunction (OBD)
Brief Title: Opioid-induced Bowel Dysfunction: Pivotal Assessment of Lubiprostone
Acronym: OPAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Sucampo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OBD0631
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2015-12

CONDITIONS: Opioid-Induced Bowel Dysfunction
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 0 mcg capsules twice daily (BID)
  Interventions: Drug: Placebo
- Lubiprostone (Experimental): 24 mcg capsules twice daily (BID)
  Interventions: Drug: Lubiprostone

INTERVENTIONS:
Drug: Lubiprostone — 24 mcg capsules twice daily (BID)
  Other Names: Amitiza®
  Arms: Lubiprostone
Drug: Placebo — 0 mcg capsules twice daily (BID)
  Other Names: No other names
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of lubiprostone administration in patients with Opioid-induced Bowel Dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Consistent treatment for chronic, non-cancer-related pain with any full agonist opioid for at least 30 days prior to screening.
* Diagnosis of opioid-induced bowel dysfunction (OBD) as confirmed during the screening period.
* If patient has a history of chronic constipation, condition must have been exacerbated by initiation of opioid treatment.
* Use of prescribed or Over-the-Counter (OTC) medication that affects gastrointestinal motility (other than opioid therapy) must be discontinued during the study.
* If treated for clinical depression with Selective serotonin reuptake inhibitor (SSRIs), Serotonin-norepinephrine reuptake inhibitor (SNRIs), or Monoamine oxidase inhibitor (MAO) inhibitors, treatment must have been at a stable dose for at least 30 days prior to screening.
* Use of laxative and stool softeners (with the exception of approved rescue medications) must be discontinued while on study.

Exclusion Criteria:

* Treatment with opioid therapy for cancer-related pain, abdominal pain, scleroderma, and/or for the management of drug addiction.
* Patient has been treated for cancer in the past 5 years (with the exception of localized basal cell, squamous cell skin cancer, or in situ cancer that has been resected).
* Opioid dose adjustment (+/- 30%), and/or change in opioid agent or route of administration within 30 days of screening.
* Gastrointestinal or abdominal surgical procedures within 90 days prior to screening.
* Non-ambulatory patients, or those who are unable to eat/drink, take oral medications, or to hold down oral medications due to vomiting.
* Female patients of childbearing potential who are unable/unwilling to use protocol-specified method(s) of birth control and/or are pregnant, nursing, or plan to become pregnant or nurse during the study.
* Prior use of Amitiza, lubiprostone, SPI-0211, or RU-0211.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (95):
- United States (94):
  - The Birmingham Pain Center, Birmingham, Alabama
  - Simon Williamson Clinic, PC, Hueytown, Alabama
  - Alabama Orthopedic Clinic, Mobile, Alabama
  - Clinical Research Advantage, Inc./ Mesa Family Medical Center, Mesa, Arizona
  - Clinical Research Advantage, Inc., Tempe, Arizona
  - Harmony Clinical Research, Inc., Tucson, Arizona
  - Verona Clinical Research, Inc., Tucson, Arizona
  - Quality of Life Medical & Research Center, LLC, Tucson, Arizona
  - Genova Clinical Research, Inc., Tucson, Arizona
  - Pusch Ridge Family Medicine / WC Clinical Research, Tucson, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Orange County Clinical Trials, Inc., Anaheim, California
  - Gregory J. Wiener, MD PC, Chula Vista, California
  - Digestive and Liver Disease Specialists, Garden Grove, California
  - RX Clinical Research, Inc, Garden Grove, California
  - Physicians Clinical Research Corporation, Laguna Hills, California
  - Loma Linda University Physicians Medical Group, Loma Linda, California
  - HealthCare Partners Medical Group, Long Beach, California
  - Impact Clinical Trials, Los Angeles, California
  - The Regents of the University of California, Los Angeles, Los Angeles, California
  - Pasadena Rehabilitation Institute, Pasadena, California
  - Northern California Research Corporation, Sacramento, California
  - SB Family Medicine, Solana Beach, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Lynn Institute of Pueblo, Pueblo, Colorado
  - Advanced Diagnostic Pain Treatment Center, New Haven, Connecticut
  - International Research Clinicians of Conneticut, Ridgefield, Connecticut
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Meridien Research, Brooksville, Florida
  - South Lake Pain Institute, Clermont, Florida
  - Century Clinical Research, Daytona Beach, Florida
  - International Medical Research, Daytona Beach, Florida
  - Clinical Physiology Associates/Clinical Study Center, Fort Myers, Florida
  - Southeaster Integrated Medical, PL d/b/a Florida Medical Research Institute, Gainesville, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - North Georgia Premier Research, Dawsonville, Georgia
  - Best Clinical Research, Decatur, Georgia
  - Drug Studies America, Marietta, Georgia
  - Pinnacle Trials Inc., Stockbridge, Georgia
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - Saltzer Medical Group, Nampa, Idaho
  - Millenium Pain Center, Bloomington, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - Redhead Research Inc., dba Research Associates of Central Illinois, Peoria, Illinois
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - The Pain Treatment Center of the Bluegrass and Ballard Wright, MD PSC, Lexington, Kentucky
  - Gulf Coast Research, LLC, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - The Willis-Knighton Pain Management Center, Shreveport, Louisiana
  - Pain and Rehabilitation Medicine, Bethesda, Maryland
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - Professional Clinical Research, Benzonia, Benzonia, Michigan
  - Center for Clinical Studies, Dearborn, Michigan
  - Apex Medical Research, AMR, Inc., Flint, Michigan
  - Digestive Health Specialists, PA, Tupelo, Mississippi
  - Impact Clinical Trials, Las Vegas, Las Vegas, Nevada
  - Office of Stephen H. Miller, MD, Las Vegas, Nevada
  - University of Nevada, Reno, Nevada
  - Cooper Health System, Camden, New Jersey
  - UMDNJ, Stratford, New Jersey
  - Partners in Primary Care, Voorhees Township, New Jersey
  - Abraham D. Morganoff, MD PA, Watchung, New Jersey
  - Northway Medical Associates, Fulton, New York
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - University of Rochester, Rochester, New York
  - Diversified Research, Durham, North Carolina
  - Medoff Medical/ Vital re:Search, Greensboro, North Carolina
  - Carolina Pharmaceutical Research, Statesville, North Carolina
  - Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Cleveland Clinic, Cleveland, Ohio
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Pain Research of Oregon, LLC, Eugene, Oregon
  - Affinity Research, Portland, Oregon
  - Private Practice of Dr. Hasan, Allentown, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Partners in Clinical Research, Cumberland, Rhode Island
  - University Gastroenterology, Providence, Rhode Island
  - Trident Institute of Medical Research, LLC, North Charleston, South Carolina
  - Southeastern Clinical Research, Chattanooga, Tennessee
  - Comprehensive Pain Specialists, PLLC, Hendersonville, Tennessee
  - Vanderbilt University - Interventional Pain Center, Nashville, Tennessee
  - Integrity Clinical Research, LLC, Savannah, Tennessee
  - Dallas VA Research Corporation, Inc., Dallas, Texas
  - Bexar Clinical Trials, LLC, Dallas, Texas
  - Permian Research Foundation, Odessa, Texas
  - Bexar Clinical Trials, LLC, Richardson, Texas
  - Salt Lake Research, PLLC, Salt Lake City, Utah
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - General Clinical Research Center, Virginia Commonwealth University, North Hospital, Richmond, Virginia
  - Metro Physicians a Division of Wheaton Franciscan Medical Group, Milwaukee, Wisconsin
  - Clement J. Zablocki VA Medical Center, Milwaukee, Wisconsin
- Health Sciences Center, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cryer B, Katz S, Vallejo R, Popescu A, Ueno R. A randomized study of lubiprostone for opioid-induced constipation in patients with chronic noncancer pain. Pain Med. 2014 Nov;15(11):1825-34. doi: 10.1111/pme.12437. Epub 2014 Apr 9. PMID 24716835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 03 August 2007 to 06 March 2009 Recruitment sites: 77 U.S. investigative sites and 3 Canadian investigative sites
Pre-assignment Details: Safety evaluable population, defined as all participants who were randomized and dosed, according to the product actually received.
Groups:
- Placebo: Placebo : 0 mcg capsules twice daily (BID) for up to 12 weeks
- Lubiprostone: Lubiprostone : 24 mcg capsules twice daily (BID) for up to 12 weeks
Period: Overall Study
Arm/Group | Placebo | Lubiprostone
Started | 218 | 221
Completed | 154 | 152
Not Completed | 64 | 69

BASELINE CHARACTERISTICS:
Population: Baseline analysis based on ITT population, which included 217 placebo-treated subjects and 221 lubiprostone-treated subjects.
Groups:
- Placebo: Placebo : 0 mcg capsules twice daily (BID)
- Lubiprostone: Lubiprostone : 24 mcg capsules twice daily (BID)
- Total: Total of all reporting groups
Arm/Group | Placebo | Lubiprostone | Total
Number analyzed (Participants) | 217 | 221 | 438
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (11.94) | 50.1 (9.89) | 50.0 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 136 | 280
  Male | 73 | 85 | 158
Region of Enrollment [Number; unit: participants]
  United States | 216 | 218 | 434
  Canada | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Weekly Spontaneous Bowel Movements at Week 8
Description: Spontaneous bowel movements (SBMs) are defined as bowel movements without the aid of drugs.
Time Frame: at Week 8
Population: Per protocol population at Week 8 without dose reduction
Measure: Mean (Standard Deviation); unit: SBMs/Week
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 169 | 164
SBMs/Week | 2.4 (3.25) | 3.2 (3.35)

2. Secondary Outcome: Mean Number of Spontaneous Bowel Movements (SBM) Per Week Within 12 Weeks
Description: Average weekly SBM frequency was calculated from data collected from Week 1 through Week 12
Time Frame: within 12 weeks
Population: Intention to treat with scores at all 12 weeks
Measure: Mean (Standard Deviation); unit: SBMs/Week
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 216 | 218
SBMs/Week
  at Week 12 | 2.2 (3.26) | 2.8 (3.60)
  within 12 weeks | 2.1 (2.35) | 2.7 (2.59)

3. Secondary Outcome: Number of Participants With the First Post-dose Spontaneous Bowel Movement Within 48 Hours Post-dose
Description: The number of participants who experienced their first post-dose Spontaneous Bowel Movement within 24 and 48 hours after dosing started.
Time Frame: within 48 hours post-dose
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 217 | 221
Participants
  within 24 hours | 65 | 89
  within 48 hours | 116 | 138

4. Secondary Outcome: Number of Participants Classified as Responders
Description: Number of participants who remained on treatment for at least 8 weeks, and reported at least 3 SBMs for at least half the weeks on study.
Time Frame: within 12 weeks
Population: Intention to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 217 | 221
Participants | 87 | 103

5. Secondary Outcome: Mean Change From Baseline in Straining, Stool Consistency, Constipation Severity, Abdominal Bloating, Abdominal Discomfort, and Bowel Habit Regularity
Description: Measures collected over 12-week treatment period were averaged, and the score at baseline was subtracted from the score at week 12 to determine the change from baseline.
  Straining scale: 0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe - higher scores are worse;
  Stool consistency scale: 0 = very loose, 1 = loose, 2 = normal, 3 = hard, 4 = very hard (little balls) - middle scores are best;
  Constipation severity scale: 0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe - higher scores are worse;
  Abdominal bloating scale: 0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe - higher scores are worse;
  Abdominal discomfort scale: 0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe - higher scores are worse;
  Bowel habit regularity scale: 7-point scale, where 1 = very regular and 7 = very irregular - higher scores are worse
Time Frame: within 12 weeks
Population: Intention to Treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 217 | 221
score on a scale
  Straining | -0.6 (0.88) | -1.0 (1.00)
  Stool consistency | -0.5 (0.77) | -0.8 (0.91)
  Constipation severity | -0.4 (0.71) | -0.6 (0.74)
  Abdominal bloating | -0.4 (0.63) | -0.4 (0.63)
  Abdominal discomfort | -0.3 (0.63) | -0.5 (0.62)
  Bowel habit regularity | -0.5 (1.63) | -0.6 (1.45)

6. Secondary Outcome: Participant Reported Outcome of Treatment Effectiveness
Description: Participants rated treatment effectiveness at the end of each treatment week during the study on a 5-point scale, where 0 = not at all effective, 1 = a little bit effective, 2 = moderately effective, 3 = quite a bit effective, 4 = extremely effective. The 12 weekly scores were averaged. Higher scores mean the drug was more effective.
Time Frame: within 12 weeks
Population: Intention to Treat with all required scores
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 214 | 211
score on a scale | 1.3 (0.99) | 1.6 (1.04)

ADVERSE EVENTS:
Time Frame: from time of first dose to 7 days after the final treatment (within 13 weeks)
Description: Treatment-emergent adverse events (TEAEs) are collected from participants based on the treatment actually received. TEAEs are defined as adverse events that began or got worse after the start of study drug. The safety evaluable population is based on the treatment actually received.
Arm/Group | Placebo | Lubiprostone
All-Cause Mortality (participants affected / at risk) | 0/218 | 0/221
Serious Adverse Events (participants affected / at risk) | 8/218 | 12/221
Other Adverse Events (participants affected / at risk) | 22/218 | 59/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=218) | Lubiprostone (N=221)
Gastroenteritis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1
Postpartum depression (Psychiatric disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Ileum fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=218) | Lubiprostone (N=221)
Nausea (Gastrointestinal disorders) | 13 | 35
Diarrhoea (Gastrointestinal disorders) | 7 | 21
Abdominal distension (Gastrointestinal disorders) | 5 | 17

LIMITATIONS AND CAVEATS:
Three participants were randomized to the wrong product, so only the safety evaluable set includes all participants according to the product actually received.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days